CLINICAL TRIAL: NCT05794178
Title: Testing Responses of Young Adults to Intervention Messages (TRY AIM) for Promoting Physical Activity Trial
Brief Title: Testing Responses of Young Adults to Intervention Messages for Promoting Physical Activity Trial
Acronym: TRY AIM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, David Conroy, Bickner Chair of Kinesiology and Professor of Kinesiology, School of Kinesiology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: STUDY00019311; R33HL164868 (NIH)
Record Dates: First submitted 2023-03-20; First posted 2023-04-03 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Physical Inactivity; Weight Gain
MeSH Terms: conditions — Sedentary Behavior; Weight Gain | interventions — Educational Status; Fitness Trackers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Precision AIM (Experimental): Education + activity monitor + up to 4 text messages/day, each drawn from one of 3 content libraries and timed based on a person- and context-specific algorithm that will be updated monthly based on incoming data (within a participant-defined availability window)
  Interventions: Behavioral: Education; Behavioral: Activity tracker; Behavioral: Text messaging (precision dosing)
- Random AIM (Active Comparator): Education + activity monitor + up to 4 text messages/day, each drawn from one of 3 content libraries and timed at random (within a participant-defined availability window).
  Interventions: Behavioral: Education; Behavioral: Activity tracker; Behavioral: Text messaging (random timing and selection)
- No AIM (Active Comparator): Education + activity monitor
  Interventions: Behavioral: Education; Behavioral: Activity tracker

INTERVENTIONS:
Behavioral: Education — Education about health benefits of physical activity, 2018 US Physical Activity Guidelines, assigned goals tailored to baseline step counts, and worksheet to develop action and coping plans (three of each)
Behavioral: Activity tracker — Fitbit activity tracker and mobile app to provide ad libitum behavioral feedback and self-regulatory support
Behavioral: Text messaging (random timing and selection) — Four text messages/day at random times within a participant's availability window and drawn at random from one of three content libraries (move more [40%], sit less [40%], inspirational quotes [20%])
  Arms: Random AIM
Behavioral: Text messaging (precision dosing) — Up to four text messages/day within a participant's availability window, timed and selected from one of three content libraries (move more, sit less, inspirational quotes) based on a person-specific dynamic model and contextual data
  Arms: Precision AIM

SUMMARY:
The goal of this clinical trial is to test a precision (person-specific and context-sensitive) messaging algorithm for increasing physical activity and slowing weight gain in insufficiently-active young adults. The main questions it aims to answer are:

* Does physical activity increase more when text messages are sent based on a precision rule for selecting and timing messages compared to when the same message content is selected and sent at random or not at all?
* Do biological or social characteristics of young adults make them more likely to respond positively to the precision messaging intervention than either of the other two interventions?

Participants will be provided with education about health-enhancing physical activity and given an activity tracker to wear for 12 months. They will then be randomly assigned to one of three groups. Participants in one group (Precision AIM) will receive up to 4 messages/day selected and timed based on a person-specific algorithm that forecasts possible message effects periodically throughout the day. Messages will be drawn from one of three content libraries: move more, sit less, or inspirational quotes. Participants in a second group (Random AIM) will receive 4 messages/day selected at random from the same three content libraries and delivered at random times within their availability window. Participants in the third group (No AIM) will receive not motivational messages but will randomly assigned to the Random AIM group will receive up to 4 messages/day drawn at random from three content libraries at randomly-selected times. Step counts and weight will be assessed at baseline, and at 3 months, 6 months, 12 months, and 18 months. Researchers will compare Precision AIM, Random AIM and No AIM groups to see if physical activity increased more and weight gain was slower in Precision AIM than Random AIM or No AIM after 3, 6, and 12 months of intervention, and 6 months after the intervention is complete (18 months).

ELIGIBILITY:
Inclusion Criteria:

* own an iPhone or Android smartphone that they would be willing to download the Fitbit app onto and sync with a Fitbit tracker and a custom, AIM app
* willing to wear a Fitbit tracker almost continually (23.5 hours/day) for a 12- month period of time
* free of visual impairment that would interfere with the receipt of text messages on their phone
* capable of reading, speaking and understanding English and of giving informed consent
* willing to complete a full 18-month study protocol

Exclusion Criteria:

* self-report sufficient aerobic activity to meet 2018 Physical Activity Guidelines for American adults
* research-grade accelerometer records sufficient aerobic physical activity to meet 2018 Physical Activity Guidelines for American adults
* living outside the continental US
* one or more contraindications to physical activity
* require an assistive device for mobility or have any other condition that may limit or prevent participation in moderate-intensity physical activity
* pregnant or planning to become pregnant within the next 12 months
* prior diagnosis of cancer, cardiovascular disease, diabetes or metabolic syndrome
* concurrent participation in another research study involving physical activity or weight loss
* planning to have surgery or relocate outside the continental US within the next year.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 360 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Average daily step counts (6 months) | Change from baseline to 6 months
  Average daily step counts recorded by Actigraph accelerometer over a 7-day monitoring period

SECONDARY OUTCOMES:
Average daily step counts (12 months) | Change from baseline to 12 months
  Average daily step counts recorded by Actigraph accelerometer over a 7-day monitoring period
Average daily step counts (18 months) | Change from 12 months to 18 months
  Average daily step counts recorded by Actigraph accelerometer over a 7-day monitoring period
Weight (6 months) | Change from baseline to 6 months
  Weight (kg) measured by BodyTrace scale
Weight (12 months) | Change from baseline to 12 months
  Weight (kg) measured by BodyTrace scale
Weight (18 months) | Change from 12 months to 18 months
  Weight (kg) measured by BodyTrace scale
Moderate-to-vigorous intensity physical activity duration (6 months) | Change from baseline to 6 months
  Average duration of daily moderate (or higher) physical activity recorded by Actigraph accelerometer over a 7-day monitoring period
Moderate-to-vigorous intensity physical activity duration (12 months) | Change from baseline to 12 months
  Average duration of daily moderate (or higher) physical activity recorded by Actigraph accelerometer over a 7-day monitoring period
Moderate-to-vigorous intensity physical activity duration (18 months) | Change from 12 months to 18 months
  Average duration of daily moderate (or higher) physical activity recorded by Actigraph accelerometer over a 7-day monitoring period
Light intensity physical activity duration (6 months) | Change from baseline to 6 months
  Average duration of daily light-intensity physical activity recorded by Actigraph accelerometer over a 7-day monitoring period
Light intensity physical activity duration (12 months) | Change from baseline to 12 months
  Average duration of daily light-intensity physical activity recorded by Actigraph accelerometer over a 7-day monitoring period
Light intensity physical activity duration (18 months) | Change from 12 months to 18 months
  Average duration of daily light-intensity physical activity recorded by Actigraph accelerometer over a 7-day monitoring period
Sedentary behavior duration (6 months) | Change from baseline to 6 months
  Average duration of daily sedentary behavior physical activity recorded by Actigraph accelerometer over a 7-day monitoring period
Sedentary behavior duration (12 months) | Change from baseline to 12 months
  Average duration of daily sedentary behavior recorded by Actigraph accelerometer over a 7-day monitoring period
Sedentary behavior duration (18 months) | Change from 12 months to 18 months
  Average duration of daily sedentary behavior recorded by Actigraph accelerometer over a 7-day monitoring period

CONTACTS AND LOCATIONS:
Overall Officials: David E Conroy, PhD, Principal Investigator — University of Michigan; Constantino M Lagoa, PhD, Principal Investigator — The Pennsylvania State University
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - The Pennsylvania State University, University Park, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided